CLINICAL TRIAL: NCT07112950
Title: The Effect of Press Needle Acupuncture on Pain Reduction and Quality of Life Improvement in Lung Cancer Patients
Brief Title: Press Needle Acupuncture for Pain and Quality of Life in Lung Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yuanti Yunus Konda, MD, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-05-0758
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer Patients

STUDY DESIGN:
Intervention Model Description: Press needle acupuncture and standart therapy will be designated as the intervention group, while the sham press needle acupucnture and standart therapy will be designated as the control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the participants and the outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The press needle acupuncture and standart therapy
  Interventions: Device: Press Needle Acupuncture and standart therapy
- Control Group (Sham Comparator): The sham press needle acupuncture and standart therapy
  Interventions: Device: Press Needle Acupuncture and standart therapy

INTERVENTIONS:
Device: Press Needle Acupuncture and standart therapy — The patient will have a press needle applied, which will be removed on the seventh day.

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of press needle acupuncture on pain management and quality of life improvement in patients with lung cancer.

The main question this study aims to answer is:

Does press needle acupuncture, when combined with standard therapy, provide better pain relief and quality of life improvement in lung cancer patients compared to standard therapy alone?

Researchers will compare press needle acupuncture to sham acupuncture to determine whether press needle acupuncture is more effective in reducing pain and improving quality of life.

Participants will:

Receive either press needle acupuncture or sham press needle acupuncture for 7 days

Visit the clinic once a week for examination and evaluation

Record improvements in pain intensity in a pain diary and assess quality of life using a quality of life questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of lung cancer through histopathology or radiology.
* Lung cancer patients aged over 18 years.
* Stage III-IV lung cancer patients receiving therapy at Dr. Cipto Mangunkusumo National General Hospital (RSUPN) and Tangerang District General Hospital (RSUD Kabupaten Tangerang).
* Patients with a VAS score >10 mm for baseline pain and >40 mm during breakthrough pain.
* Willing to participate in the study until completion by signing the informed consent form.

Exclusion Criteria:

* Lung cancer patients with deteriorating general condition.
* Presence of wounds or infections at the press needle insertion site.
* History of allergy to stainless steel materials.
* Patients with blood clotting disorders: platelet count <50,000/μL, ANC <1000/mm³, or patients undergoing anticoagulant therapy with INR >2.142.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for Pain | Before therapy, Day 1, Day 3, Day 7, and Day 14
  Pain intensity will be measured using the Visual Analogue Scale (VAS), which consists of a horizontal or vertical line 10 cm (100 mm) in length, representing a continuum of pain intensity from:
  0 = No pain at all
  10 = Worst imaginable pain

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Lung (FACT-L) | Before therapy, Day 7, and Day 14
  Quality of life will be assessed using the FACT-L questionnaire, consisting of 37 items rated on a 0-4 Likert scale:
  0 = Not at all
  1. = A little bit
  2. = Somewhat
  3. = Quite a bit
  4. = Very much
  Total scores range from 0 to 28 (higher scores indicate better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee of Faculty of Medicine
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No